CLINICAL TRIAL: NCT01937936
Title: Stress and Health in Family Caregivers of Persons With Heart Failure
Brief Title: Heart Failure Caregiver Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Boyoung Hwang, PhD, RN, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5K23NR013475 (NIH); 5K23NR013475 (NIH)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Stress; Depression
Keywords: caregiver stress; depression; quality of life; cognitive behavioral therapy
MeSH Terms: conditions — Depression; Caregiver Burden | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Education (Active Comparator): Health Education
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Family caregivers in the CBT group will receive 8 1-hour weekly Cognitive Behavioral Therapy (CBT) sessions, which will take place in their home.
  Other Names: Cognitive Therapy; Cognitive Behavioral Intervention; CBT
  Arms: CBT
Behavioral: Health Education — Family caregivers in the Education group will receive 8 1-hour weekly sessions of general health education on selected topics, which will take place in their home.
  Arms: Education

SUMMARY:
Family caregivers are vulnerable to health problems because of the stress and demands of their role as a caregiver. With the growing incidence of heart failure (HF) and the anticipated growth in the aging population, the number of HF caregivers is expected to rise. This study will pilot test a cognitive behavioral intervention designed to reduce stress among HF caregivers, which will ultimately contribute to promoting health and quality of life among HF caregivers and their loved ones with HF.

ELIGIBILITY:
Patient Inclusion Criteria:

* 21 years or older
* Having primary or secondary diagnosis of HF (NYHA class II-IV)
* Having a family member or friend providing care for them at home
* Being able to communicate in English

Patient Exclusion Criteria:

* Being on the transplant list
* Having terminal illness (e.g., terminal cancer)

Caregiver Inclusion Criteria:

* 21 years or older
* Having the primary responsibility for the care of the patient for at least 6 months
* Living in the greater Los Angeles area
* Being able to communicate in English

Caregiver Exclusion Criteria:

* Being a paid caregiver (an individual who is hired to provide care for the patient)
* Having terminal illness (e.g., terminal cancer) or a serious medical condition that requires ongoing medical care (e.g., cancer requiring ongoing chemotherapy or radiation therapy)
* Having a history of major psychiatric illness (i.e., schizophrenia, bipolar disorder, and/or any personality disorder)
* Diagnosed with Cushing's or Addison's disease
* Taking medication that could influence cortisol levels (e.g., steroid based anti-inflammatory drugs)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | 8 weeks

SECONDARY OUTCOMES:
Perceived stress | 8 weeks and 6 months
Depressive symptoms | 8 weeks and 6 months
Health-related quality of life | 8 weeks and 6 months
Health care usage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boyoung Hwang, PhD, RN, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California

REFERENCES:
- [Derived] Hwang B, Granger DA, Brecht ML, Doering LV. Cognitive behavioral therapy versus general health education for family caregivers of individuals with heart failure: a pilot randomized controlled trial. BMC Geriatr. 2022 Apr 5;22(1):281. doi: 10.1186/s12877-022-02996-7. PMID 35382758